CLINICAL TRIAL: NCT04328545
Title: Transcranial Direct Current Stimulation Effect on Pain Threshold and Working Memory in Healthy Adolescents, Young Adults and Elderly: a Randomized , Cross-over, Single Blind Trial
Brief Title: Transcranial Direct Current Stimulation Effect on Pain Threshold and Working Memory: Impact of Age and Protocol Type
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0188
Record Dates: First submitted 2019-10-31; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Transcranial Direct Current Stimulation; Working Memory; Pain
Keywords: Age Groups; Pain Threshold
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: single (participants)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS on DLPFC (Experimental): Participants will receive anodal tDCS on the left DLPFC for 30 mins duration, cathode will be placed over the right supra orbital area. The electrodes are 25cm², The stimulation current is 2 milliamperes (2mA).
  Interventions: Device: Anodal tDCS on DLPFC
- Anodal tDCS on M1 (Active Comparator): Participants will receive anodal tDCS on the left M1 for 30 min duration, cathode will be placed over the right supra orbital area. The electrodes are 25cm², The stimulation current is 2 milliamperes (2mA).
  Interventions: Device: Anodal tDCS on M1
- Sham tDCS (Sham Comparator): Participants will receive sham tDCS. The anode will be placed on the left DLPFC and the cathode on the over the right supra orbital area. The electrodes are 25cm², There will be a ram up and down of 30 seconds each, after the ramp up the current will be turned off.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Anodal tDCS on DLPFC — Participants will receive anodal tDCS on the left DLPFC for 30 min duration, cathode will be placed over the right supra orbital area. The electrodes are 25cm², The stimulation current is 2 milliamperes (2mA).
  Other Names: DLPFC
  Arms: Anodal tDCS on DLPFC
Device: Anodal tDCS on M1 — Participants will receive anodal tDCS on the left M1 for 30 min duration, cathode will be placed over the right supra orbital area. The electrodes are 25cm², The stimulation current is 2 milliamperes (2mA).
  Other Names: M1
  Arms: Anodal tDCS on M1
Device: Sham tDCS — Participants will receive sham tDCS. The anode will be placed on the left DLPFC and the cathode on the over the right supra orbital area. The electrodes are 25cm², There will be a ram up and down of 30 seconds each, after the ramp up the current will be turned off.
  Other Names: Sham
  Arms: Sham tDCS

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive neuromodulation method which has great potential as an aid in the therapeutic management of neuropsychiatric disorders and chronic pain syndromes. However, despite promising results, the response to stimulation presents great variability among subjects. Age is a factor that is known to influence the tDCS effect forging the inconsistency of clinical effect.The purpose of this study is to evaluate the effect of tDCS on pain perception and working memory in healthy women from 3 different age groups: adolescents, young adults and elderly. This is a randomized, single-blinded, cross-over study of 2 different active interventions and sham.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a neuromodulation method that has great potential as an aid in the therapeutic management of neuropsychiatric disorders and chronic pain syndromes. tDCS modulates the neuronal membrane potential , facilitating neuronal depolarization or hyperpolarization, hence modifying the cortical excitability of the stimulated area. However, despite promising results the response to stimulation presents great variability among subjects. Chronological age is an important factor in the variation of brain plasticity. The dorsolateral prefrontal cortex (DLPFC) is associated with cognitive and emotional aspects of pain, in addition to being related to executive components of working memory. Anodal tDCS on DLPFC modulates pain level in patients with chronic pain and modifies working memory performance in healthy subjects and patients with memory impairment. The prefrontal cortex presents a great structural difference throughout lifespan: it is under maturational process in the adolescence, reaching peak of maturation in the adult life, and initiating process of cerebral senescence in elderly subjects. Therefore, the use of tDCS on DLPFC in these three age groups presents potential for a large variation in response. Faced with the potential of tDCS for adjuvant use in the treatment of several diseases, it is imperative to understand the variability of this intervention between different age groups. This knowledge may allow the optimization of neuromodulation protocols, allowing more careful and refined use in the clinic. The study primary outcomes is the difference between and within age groups on the variation of pre and post tDCS on pain threshold evaluated by Heath pain threshold on a Quantitative sensory testing paradigm and working memory performance evaluated by n-back test in healthy subjects of three age groups: adolescents, young adults, elderly. This is a randomized, single blinded, cross-over, sham-controlled clinical trial. The study will be conducted at the Clinical Research Center of the Hospital de Clínicas of Porto Alegre (HCPA). It will include 30 women, 10 women by age group: adolescents between 15 and 16 years,young adults between 30 and 40 years old and elderly women between 60 and 70 years. Participants will be randomized for a cross-over of three sessions: anodal stimulation in DLPFC, anodal stimulation in primary motor cortex (M1) as active control and sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 to 16 years for the adolescent group
* Age between 30 to 40 years for the young adult group
* Age between 60 to 70 years for the elderly group
* From completed elementary school to incomplete superior education
* right handed

Exclusion Criteria:

* Pregnancy
* Current smoker or previous smoker within 10 years
* Current Substance Use Disorder
* Neurological condition (e.g., traumatic brain injury, stroke, brain tumor, epilepsy, brain surgery, brain implant)
* Any diagnosed Psychiatric condition (e.g., Attention deficit/hyperactivity deficit (ADHD), bipolar disorder, major depressive disorder, schizophrenia, generalized anxiety disorder)
* Use of any antidepressive or psychoactive, psychostimulant medication
* Any chronic pain condition

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Heat pain Threshold | percentual change from before the tDCS onset, to immediately after the end of tDCS application for each cross-over session
  Using the Quantitative sensory testing, this measure consists of the average temperature of 3 stimulus with increasing magnitude of heat where the participant presses a button to indicate when he/she first perceives pain.
Working memory performance | up to 60 minutes after tDCS onset
  Working memory performance will be evaluated by a computerized n-back test associated with flankers at baseline and after each session of active tDCS (DLPFC or M1) or sham. The measure of performance is the D' discrimination index (calculated based on hit rate and false alarm rate).

SECONDARY OUTCOMES:
Inhibitory control performance | up to 60 minutes after tDCS onset
  A computerized stop-signal task associated with flankers will evaluate inhibitory control. Performance index are calculated with the D' discrimination index (based on hits and false alarms for go and stop trials). The task will be performed at baseline and after the stimulation on each cross-over session.
Area under the curve of the ERP during inhibitory control task | up to 60 minutes after tDCS onset
  Area under the curve of the signal of event-related potential (ERP) evoked during the stop signal task with flankers (inhibitory control performance). The signal will be assessed using an 8 channel EEG device at baseline and after each cross-over session.
Heat thermal threshold | percentual change from before the tDCS onset, to immediately after the end of tDCS application for each cross-over session
  Using the Quantitative sensory testing, this measure consists of the average temperature of 3 stimulus with increasing magnitude of heat where the participant presses a button to indicate when he/she first perceives heat.
Heat pain tolerance | percentual change from before the tDCS onset, to immediately after the end of tDCS application for each cross-over session
  Using the Quantitative sensory testing, this measure consists of the temperature for a stimulus with increasing magnitude of heat where the participant presses a button to indicate the maximum heat tolerated.
Moderate pain | percentual change from before the tDCS onset, to immediately after the end of tDCS application for each cross-over session
  Using the Quantitative sensory testing, this measure consists of the average temperature of 3 stimulus with increasing magnitude of heat where the participant presses a button to indicate pain perceived at a moderate level, i.e. level of 6 in a numeric pain scale (0 to 10).
Unpleasantness sensation | percentual change from before the tDCS onset, to immediately after the end of tDCS application for each cross-over session
  This measure will be assessed using a numeric pain scale (0 to 10 in which 0 represents no unpleasant sensation and 10 extremely unpleasant sensation) with which participant will indicate how unpleasant was the temperature of the quantitative sensory testing stimulus for the heat pain threshold.
Alpha wave power | up to 60 minutes after tDCS onset
  Assessment of alpha wave power (8Hz to 12Hz) will be done using an 8 channel EEG device during an "eyes-open and eyes-closed" paradigm where participant is in a resting state at baseline and after each cross-over session.
Beta wave power | up to 60 minutes after tDCS onset
  Assessment of beta wave power (12Hz to 25Hz) will be done using an 8 channel EEG device during an "eyes-open and eyes-closed" paradigm where participant is in a resting state at baseline and after each cross-over session.
Theta wave power | up to 60 minutes after tDCS onset
  Assessment of theta wave power (4Hz to 8Hz) will be done using an 8 channel EEG device during an "eyes-open and eyes-closed" paradigm where participant is in a resting state at baseline and after each cross-over session.
serum BDNF levels | up to 60 minutes before tDCS onset
  Neuroplasticity biomarker will be assessed using serum brain-derived neurotrophic factor (BDNF) at baseline to be correlated with tdcs effects on primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with coded variables and coded participant numbers, only to editors and reviewers of journals where the studies are submitted and registered and under formal request
Supporting Information: Study Protocol, ICF
Time Frame: Available in August 2019; Available for 3 years
Access Criteria: by e-mail, under request

REFERENCES:
- [Background] Gazzaley A, Cooney JW, Rissman J, D'Esposito M. Top-down suppression deficit underlies working memory impairment in normal aging. Nat Neurosci. 2005 Oct;8(10):1298-300. doi: 10.1038/nn1543. Epub 2005 Sep 11. PMID 16158065
- [Background] Palm U, Segmiller FM, Epple AN, Freisleder FJ, Koutsouleris N, Schulte-Korne G, Padberg F. Transcranial direct current stimulation in children and adolescents: a comprehensive review. J Neural Transm (Vienna). 2016 Oct;123(10):1219-34. doi: 10.1007/s00702-016-1572-z. Epub 2016 May 12. PMID 27173384
- [Background] Scharinger C, Soutschek A, Schubert T, Gerjets P. When flanker meets the n-back: What EEG and pupil dilation data reveal about the interplay between the two central-executive working memory functions inhibition and updating. Psychophysiology. 2015 Oct;52(10):1293-304. doi: 10.1111/psyp.12500. Epub 2015 Aug 3. PMID 26238380
- [Result] Boggio PS, Zaghi S, Lopes M, Fregni F. Modulatory effects of anodal transcranial direct current stimulation on perception and pain thresholds in healthy volunteers. Eur J Neurol. 2008 Oct;15(10):1124-30. doi: 10.1111/j.1468-1331.2008.02270.x. Epub 2008 Aug 20. PMID 18717717
- [Result] Fregni F, Boggio PS, Nitsche M, Bermpohl F, Antal A, Feredoes E, Marcolin MA, Rigonatti SP, Silva MT, Paulus W, Pascual-Leone A. Anodal transcranial direct current stimulation of prefrontal cortex enhances working memory. Exp Brain Res. 2005 Sep;166(1):23-30. doi: 10.1007/s00221-005-2334-6. Epub 2005 Jul 6. PMID 15999258
- [Derived] Saldanha JS, Zortea M, Deliberali CB, Nitsche MA, Kuo MF, Torres ILDS, Fregni F, Caumo W. Impact of Age on tDCS Effects on Pain Threshold and Working Memory: Results of a Proof of Concept Cross-Over Randomized Controlled Study. Front Aging Neurosci. 2020 Jun 30;12:189. doi: 10.3389/fnagi.2020.00189. eCollection 2020. PMID 32714178